CLINICAL TRIAL: NCT02447042
Title: Study of Changes on Mean Systemic Filling Pressure (Pmsf) and Microcirculation After a Fluid Challenge in Septic Patients: Looking for the Minimal Volume
Brief Title: Minimal Volume for a Fluid Challenge in Septic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Principal Investigator, HollmannAya, Research Fellow Intensive Care Directorate, St George's, University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14.0156
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Sepsis
Keywords: sepsis; Fluids; Mean systemic filling pressure
MeSH Terms: conditions — Sepsis | interventions — Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 ml/Kg (Experimental): Fluid challenge with crystalloids (2 ml/Kg) infused in 5 minutes Measurment of Pmsf-arm before and after the fluid challenge
  Interventions: Procedure: Fluid challenge with crystalloids; Device: Measurement of Pmsf-arm
- 3 ml/Kg (Experimental): Fluid challenge with crystalloids (3 ml/Kg) infused in 5 minutes Measurment of Pmsf-arm before and after the fluid challenge
  Interventions: Procedure: Fluid challenge with crystalloids; Device: Measurement of Pmsf-arm
- 4 ml/kg (Experimental): Fluid challenge with crystalloids (4 ml/Kg) infused in 5 minutes Measurment of Pmsf-arm before and after the fluid challenge
  Interventions: Procedure: Fluid challenge with crystalloids; Device: Measurement of Pmsf-arm
- 5 ml/Kg (Experimental): Fluid challenge with crystalloids (5 ml/Kg) infused in 5 minutes Measurment of Pmsf-arm before and after the fluid challenge
  Interventions: Procedure: Fluid challenge with crystalloids; Device: Measurement of Pmsf-arm

INTERVENTIONS:
Procedure: Fluid challenge with crystalloids — Intravenous infusion of 2, 3, 4 or 5 ml/Kg of crystalloids over 5 minutes.
Device: Measurement of Pmsf-arm — Measurement of stop-flow arterial-venous equilibrium pressure in the arm where the radial arterial pressure is measured by inflating a pneumatic cuff with an automatic pneumatic tourniquet during 60 seconds before and after the fluid challenge in patients receiving 2 ml/Kg, 3 ml/kg, 4 ml/kg and 5 ml/kg of crystalloids in 5 minutes
  Other Names: Meassurement of mean systemic filling pressure - arm

SUMMARY:
The administration of fluids intravenously is the first step in the stabilization of patients in septic shock. It is important to give the right dose of fluids, enough to improve the function of the cardiovascular system but not too much to drown the cells in water. In order to know that, the investigators use the "fluid challenge" which is the administration of a "small amount" of fluid in a short period of time in order to test the cardiovascular response to a dose of fluids. However, it is unclear how "small" this amount can be. The aim of this study is to find out the minimum volume required to perform an effective "fluid challenge". The investigators hypothesize that the changes in the mean pressure in the cardiovascular system (socalled mean systemic filling pressure or Pmsf) during the administration of small amounts of fluid can be used to detect the minimum volume required to effectively test the cardiovascular system with a fluid challenge.

On the other hand, microcirculation may remain impaired despite the stabilization of the macrocirculation. The microcirculation can be much more dynamic than the macrocriculation, so it is essential to observe the changes of both over time. Patients admitted at the investigators' intensive care unit (ICU) due to sepsis can be included in this study. The sample will be divided in 4 groups according to the volume of the fluid challenge: 2 ml/kg, 3 ml/kg, 4ml/Kg and 5 ml/kg.

The investigators will measure the Pmsf non-invasively using a pneumatic tourniquet inflated during one minute. Invasive arterial blood pressure will be observed during the inflation of the cuff in the arm to determine the Pmsf. The least significant change of Pmsf using this method is 14%. The minimal volume will be that one that achieve that change in Pmsf.

DETAILED DESCRIPTION:
PURPOSE AND DESIGN The main objective of this study is to find out the minimum volume of fluid required to perform an effective "fluid challenge" in septic patients. An effective fluid challenge would be one that is able to increase the mean pressure in the cardiovascular system when there is no blood circulation or socalled the mean systemic filling pressure (Pmsf). It is similar to the pressure into a pneumatic tyre, which is only related to the volume of air and the elastic properties of the tyre wall. In order to do this, the investigators will observe the changes in mean systemic filling pressure after small amounts of fluids so that the investigators will be able to realise how much volume is required to increase that pressure.

To assure that the change in Pmsf is a real change, the investigators have conducted a pilot study in order to determine the precision of the Pmsf measurement using the Pmsf-arm technique. The least significant change is about 14 % from baseline measurement. The Pmsf-arm technique is a process very similar to that the investigators use to measure non-invasive blood pressure. The investigators will measure the arterial-venous equilibrium pressure in the arm after a rapid and brief interruption of blood circulation. In order to do this, a totally noninvasive automatic tourniquet is attached to the arm where the arterial line has been inserted and the tourniquet is inflated during 60 seconds. This process will be done at baseline and after the fluid challenge. The second objective is observe the microcirculation during an affective fluid challenge and correlate the changes observed with the changes in the cardiac function and the Pmsf.

The third objective is to observe the changes generated by the vasoactive therapy in the macro and microcirculation according to the cardiac response and the type of vasoactive therapy used.

In the investigators' clinical practice, the investigators have observed that in some cases the infusion of 250 ml of fluid has no impact at all in the cardiovascular function. The investigators believe that in those cases the investigators may have not given enough fluid to increase the Pmsf and test the cardiovascular response.

RECRUITMENT The sample will be recruited by convenience. It is important to understand the difference between fluid resuscitation and fluid challenge. The fluid resuscitation requires normally large amount of volume in a medical emergency in order to achieve cardiovascular stability. Once the patient is minimally stable, a fluid challenge is normally carried out in order to find out if the patient may benefit from more fluids. As the performance of a fluid challenge is part of the normal clinical practice once the patient has been admitted to ICU, there is minimal extra risk from participation in this study.

CONSENT Informed consent will be required to become participant of this study. Informed consent will be obtained by the Principal Investigator who has also clinical responsibility for the care of patients under the care of the intensive care department. The PI has received training in Good Clinical Practice (GCP).

RISK, BURDENS AND BENEFITS Currently, the investigators use a fluid administration protocol in septic patients based on the principle of "stroke volume maximization". The investigators perform a fluid challenge of about 4 ml/kg until the patient becomes "non-responder", which means that the heart is not able to increase the volume ejected anymore. However, the investigators have observed some pitfalls in this protocol. Some patients classified as "non-responders" may need more than 4 ml/kg to test the cardiovascular response. The investigators' hypothesis is that in those cases, the cardiovascular system is either very relaxed or very empty, and 4 ml/kg was not enough to increase the mean systemic filling pressure. Therefore, a possible benefit associated to this study is to avoid this possible pitfall. If after a fluid challenge the Pmsf has not changed significantly, the clinician in charge will be informed and he/she will decide whether continue with a subsequent fluid challenge until the investigators observe a significant change on Pmsf.

There are not relevant risk from participation in the study. As fluid challenge will be performed in accordance with the clinician prescription, the observations are non-invasive and do not involve any risk for the participant and arterial line is normally used in these patients, there is minimal extra risk from participating in this study.

CONFIDENTIALITY Identifiable data will not be obtained for the purpose of this study. All the data (case report forms and electronic files) will be anonymised. The participant will be identified with a code that will be generated specifically for this study.

The "identification code" generated for the participant will be linked to the "hospital number" and to the name of the patient, by a secret rule that is kept confidentially by the principal researcher. This rule will only be used in case of missing information that can be completed retrospectively. The only person able to access to identifiable information is the principal investigator, who is aware of the responsibility of the confidentiality of this study.

All the data collected will be stored in encrypted electronic memories and the written material in custody of the principal investigator. No written material will contain identifiable data.

CONFLICT OF INTEREST During the period of study, the principal investigator will not be responsible for the participant's care at the same time, in order to avoid conflict of interest. However, the principal investigator retains clinical responsibility for the care of patients as member of the intensive care department.

At the end of the study, the investigators are planning to use this information as a chapter for a doctoral thesis, to present the study in international conferences and, hopefully, to publish the results in scientific journals.

If the patient wishes to be informed of the results of this study, the investigators will send a copy of the abstract presented in international conferences by email, or a copy of the paper accepted in a medical journal by email.

ELIGIBILITY:
Inclusion Criteria:

Fulfil 2 of 4 of the criteria of the systemic inflammatory response syndrome (SIRS) due to known or suspected infection within the previous 24 hours. The SIRS criteria are:

1. Core temperature >38 °C or < 36 °C
2. Tachycardia (heart rate > 90 beats per minute)
3. Tachypnoea (respiratory rate >20 breaths per minute or PaCO2 < 4.3 kPa or need for mechanical ventilation)
4. Abnormal white cell count (> 12000 cells/mm3 or < 4000 cells/mm3, or >10% immature (band cells) forms.

Exclusion Criteria:

* Extensive peripheral arterial occlusive disease in upper limbs.
* Postoperative valvular insufficiency
* Aortic valve regurgitation
* Tachyarrhythmia
* Cardiac assist device (IntraAortic balloon pump)
* Previously known right ventricular failure
* Known vasospastic diseases, systemic sclerosis or Raynaud's phenomenon.
* Patients requiring aggressive fluid resuscitation due to lifethreatening cardiovascular instability
* Known pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Pmsf-arm (expressed in percentage from baseline value) | Inmediately after end of fluid infussion

SECONDARY OUTCOMES:
Change in cardiac output (expressed in percentage from baseline value | Inmmediately after end of fluid infussion
Proportion of responders in each group | As average three moths after end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hollmann D Aya, MD, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (1):
- St George's University Hospitals, NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GUYTON AC. Determination of cardiac output by equating venous return curves with cardiac response curves. Physiol Rev. 1955 Jan;35(1):123-9. doi: 10.1152/physrev.1955.35.1.123. No abstract available. PMID 14356924
- [Background] Pinsky MR. Instantaneous venous return curves in an intact canine preparation. J Appl Physiol Respir Environ Exerc Physiol. 1984 Mar;56(3):765-71. doi: 10.1152/jappl.1984.56.3.765. PMID 6368503
- [Background] Maas JJ, Geerts BF, van den Berg PC, Pinsky MR, Jansen JR. Assessment of venous return curve and mean systemic filling pressure in postoperative cardiac surgery patients. Crit Care Med. 2009 Mar;37(3):912-8. doi: 10.1097/CCM.0b013e3181961481. PMID 19237896